CLINICAL TRIAL: NCT05064566
Title: Clinical Performance of Diagnostic Methods in Early Occlusal Caries
Brief Title: Evaluation of Caries Detection Methods
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nazan Kocak Topbas (Other)
Collaborators: Mersin University (Other)
Responsible Party: Sponsor-Investigator, Nazan Kocak Topbas, Assist. Prof. Dr., Mersin University
Organization: Mersin University (Other)
Other Study IDs: 2017-1-AP1-2000
Record Dates: First submitted 2021-05-28; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Caries; Diagnoses Disease
Keywords: Caries detection;; laser fluorescence; micro-CT; visual analog scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- caries diagnosis: diagnostic accuracy of clinical visual examination (ICDAS II), digital intraoral radiography, near infrared light transillumination (NIR-LT), and laser fluorescence (LF), by examining third molar teeth in comparison to gold standard micro-CT images.
  Interventions: Device: caries assessment

INTERVENTIONS:
Device: caries assessment — clinical visual examination (ICDAS II), digital io radiography, near infrared light transillumination (NIR-LT), and laser fluorescence (LF), and micro-CT images.

SUMMARY:
The investigators aim will be to compare the diagnostic performance of clinical visual examination (ICDAS II), intraoral/bite wing radiography (BW), near infrared light transillumination (NIR-LT), and laser fluorescence (LF), in comparison to microcomputed tomography (micro-CT) for the detection of non-cavitated occlusal enamel and dentin caries in third molar teeth. Potential participants will be consecutively recruited.

DETAILED DESCRIPTION:
Studies regarding comparison of diagnostic techniques for caries detection are generally conducted under in vitro conditions due to ethical concerns. Considering the many recently published in vitro studies which attempted to assess the diagnostic ability of different caries diagnosis systems, it is not possible to know at what rate in vitro findings are applicable to the clinical situation.The investigators would like to assess initial occlusal caries lesions by using different diagnostic methods under in vivo conditions. In the present study, the investigators will assess diagnostic accuracy of clinical visual examination (ICDAS II), digital intraoral radiography, near infrared light transillumination (NIR-LT), and laser fluorescence (LF), by examining third molar teeth in comparison to gold standard micro-CT images. The null hypothesis of the study is that no significant difference exists for the clinical performance of the evaluated methods in detecting non-cavitated occlusal caries in either the enamel or the dentin. This prospective study will include 101 third molars of 101 patients with non-cavitated occlusal caries requiring extraction. ICDAS II, BW, NIR-LT and LF examinations will be carried out by two examiners. Gold standard will be determined by micro-CT imaging after extraction. Intraclass correlation coefficient (ICC) value will be calculated for examiner agreement. Accuracy rate, sensitivity, specificity, predictive values and areas under receiver operating characteristic curves (Az) will be calculated. Clinical application time and patient comfort/pain analysis will be compared. Nonparametric variables will be assessed by Kruskal Wallis Test. Significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* According to the American Society of Anesthesiologists (ASA) only status 1/ healthy patients
* Completely erupted permanent dentition,
* No fixed orthodontic apparatus, prosthetic restoration and filling material,
* A minimum age of 18 years,
* At least one third erupted molar teeth (third mandibular or third maxillary molar from each patient was included),
* Non cavitated occlusal caries,
* Teeth with no hypoplasia or hypomineralization,
* Third molar teeth that require extraction for surgery, orthodontics and prosthetic reasons,
* If clinical indicators suggest a current caries risk or activity that required additional diagnosis, the patients will be asked to participate in this additional examination.

Exclusion Criteria:

* Patients younger than 18
* Patients that can not be recruited according to the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample will be comprised of 100 third molars requiring extraction with non-cavitated but suspected occlusal caries from 101 patients.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 1 month
  The accuracy of caries detection methods will be evaluated when compared to the gold standard Micro CT.
Receptor operating characteristic (ROC) curves | 1 month
  Receptor operating characteristic (ROC) curves (Az) will be calculated to show the caries distinguishing ability of each caries detection method and the observer.
Intraclass correlation coefficient (ICC) | 1 month
  Intra- and inter-observer reproducibility will be assessed by intraclass correlation coefficient (ICC).

SECONDARY OUTCOMES:
Patient comfort/pain analysis by using Visual Analog Scale (VAS)(comparative assessment of the tests): | 1 month
  The patients will be asked to rate their feelings (based on comfort and pain) from absence of discomfort and pain to extreme discomfort and pain (between 0 and 10) for each clinical method.
Clinical time efficacy (comparative assessment of the tests) | 1 month
  Clinical application times from the beginning of the procedure to the end of the procedure for each method will be calculated by using a stopwatch. (example: LF pen 10 sn)

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Koçak Topbaş, PhD, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)